CLINICAL TRIAL: NCT01684553
Title: The Effect of Changing the Eating Speed on Energy Intake: a Randomized Cross-over Study
Brief Title: The Effect of Changing the Eating Speed on Energy Intake
Acronym: EatSpeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Meena Shah, Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: F10-39
Record Dates: First submitted 2012-09-05; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Oral Intake Reduced
Keywords: Eating speed; energy intake

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow eating condition (Experimental): The subjects were asked to eat their meal slowly during the slow eating condition
  Interventions: Behavioral: Slow eating condition
- Fast eating condition (Active Comparator): The subjects were asked to eat their meal quickly during the fast eating condition
  Interventions: Behavioral: Fast eating condition

INTERVENTIONS:
Behavioral: Slow eating condition — The subjects were asked to eat their meal slowly during the slow eating condition
  Arms: Slow eating condition
Behavioral: Fast eating condition — The subjects were asked to eat their meal quickly during the fast eating condition
  Arms: Fast eating condition

SUMMARY:
It was hypothesized that eating a meal slowly would lead to a lower meal energy intake and lesser feelings of hunger and desire to eat and higher levels of fullness after the meal compared to eating the same meal more quickly.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 19-65 years.

Exclusion Criteria:

* Severe obesity (BMI ≥ 40 kg/m2),
* dieting,
* taking medications that affect appetite,
* participating in > 150 min/wk of vigorous physical activity,
* smoking,
* drinking heavily (men: > 14 alcoholic drinks/wk; women: > 7 alcoholic drinks/wk),
* self-reported disordered eating,
* depression,
* type 1 or 2 diabetes,
* adrenal disease, or
* untreated thyroid disease.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Meal energy intake | Day 1
Meal energy intake | Day 2

SECONDARY OUTCOMES:
Hunger questionnaire | 0 and 60 min after the meal began
Fullness questionnaire | 0 and 60 min after the meal began
Desire to eat questionnaire | 0 and 60 min after the meal began
Thirst questionnaire | 0 and 60 min after the meal began

CONTACTS AND LOCATIONS:
Overall Officials: Meena Shah, Ph.D., Principal Investigator — Tzu Chi University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States